CLINICAL TRIAL: NCT05591807
Title: Investigation to the Mechanism of the Neuroplastic Modulation in Central Auditory Tract by Electroacupuncture and Its Clinical Therapeutic Implications
Brief Title: Investigation to the Mechanism of the Neuroplastic Modulation in Central Auditory Tract
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH103-REC2-149(CR-3)
Record Dates: First submitted 2022-09-13; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Tinnitus; Neuromodulation; Electroacupuncture; Cochlear Diseases; Therapy
MeSH Terms: conditions — Tinnitus; Cochlear Diseases | interventions — Electroacupuncture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Other: Electroacupuncture — insert the acupuncture needle to SJ3(left side) and connect the electroacupuncture device for 15min, 2mA and 2Hz

SUMMARY:
Tinnitus is the awareness of sound or noise in the absence of acoustic stimulation. No definite therapeutic strategy of tinnitus has been developed yet. The current theory of tinnitus is the plasticity theory of neurophysiology model. Although acupuncture has its role in tinnitus treatment, its actual role still remains to be elucidated. Acupuncture has been proposed to induce the development of neuroplasticity. The aim of this project is to undergo a comprehensive investigation to the central auditory effect and the therapeutic effects of acupuncture in tinnitus. According the results of the preliminary studies, the objective auditory measurement and subjective tinnitus perception will be analyzed in tinnitus patients before and after acupuncture.

DETAILED DESCRIPTION:
Hearing loss is a common sensory deficit in human beings. Besides communication handicaps, hearing loss may associate with niggling tinnitus symptoms. Tinnitus is the awareness of sound or noise in the absence of acoustic stimulation. Tinnitus may cause bothersome problems in cognition, mood, or psychosocial behaviour and constitute a significant portion in the outpatient clinics of ENT practice. No definite therapeutic strategy of tinnitus has been developed yet. The current theory of tinnitus is the plasticity theory of neurophysiology model. According to this theory, several neuromodulation methods have been proposed such as repetitive transcranial magnetic stimulation (rTMS) or vagus nerve stimulation (VNS). Although acupuncture has its role in tinnitus treatment, its actual role still remains to be elucidated. Acupuncture has been proposed to induce the development of neuroplasticity. There are still few thorough researches to investigate the neurophysiological events after acupuncture. The aim of this project is to undergo a comprehensive investigation to the central auditory effect and the therapeutic effects of acupuncture in tinnitus. According the results of the preliminary studies, the objective auditory measurement and subjective tinn itus perception will be analyzed in tinnitus patients before and after acupuncture. The ultimate results of this project will clarify the basic central auditory effects of acupuncture and provide a potential for translational application of acupuncture to treat the common tinnitus patients.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 y/o
* Normal hearing
* No acupuncture contraindication

Exclusion Criteria:

* Heart disease or other acupuncture contraindication
* Bleeding tendency
* Autoimmune disease
* Drug abuse
* Pregnant or breast-feeding
* Hearing loss
* Active otitis media or inner ear diseases or retro-cochlear pathology
* Incomplete treatment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal population
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2019-07-24 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Auditory brainstem response Wave I, III and V latency | Day 0
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Auditory brainstem response Wave I, III and V amplitude | Day 0
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Auditory brainstem response Wave I, III and V latency | After electroacupuncture(Day 7)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Auditory brainstem response Wave I, III and V amplitude | After electroacupuncture(Day 7)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Auditory brainstem response Wave I, III and V latency | 7 days after electroacupuncture(Day 14)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Auditory brainstem response Wave I, III and V amplitude | 7 days after electroacupuncture(Day 14)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Middle latency response wave Na, Pa, Nb, Pb latency | Day 0
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Middle latency response wave Na, Pa, Nb, Pb amplitude | Day 0
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Middle latency response wave Na, Pa, Nb, Pb latency | After electroacupuncture(Day 7)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Middle latency response wave Na, Pa, Nb, Pb amplitude | After electroacupuncture(Day 7)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Middle latency response wave Na, Pa, Nb, Pb latency | 7 days after electroacupuncture(Day 14)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Middle latency response wave Na, Pa, Nb, Pb amplitude | 7 days after electroacupuncture(Day 14)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Late latency response wave P1, N1, P2, N2 latency | Day 0
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Late latency response wave P1, N1, P2, N2 amplitude | Day 0
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Late latency response wave P1, N1, P2, N2 latency | After electroacupuncture(Day 7)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Late latency response wave P1, N1, P2, N2 amplitude | After electroacupuncture(Day 7)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Late latency response wave P1, N1, P2, N2 latency | 7 days after electroacupuncture(Day 14)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
Late latency response wave P1, N1, P2, N2 amplitude | 7 days after electroacupuncture(Day 14)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
p300 cortical response wave latency | Day 0
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
p300 cortical response wave amplitude | Day 0
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
p300 cortical response wave latency | After electroacupuncture(Day 7)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
p300 cortical response wave amplitude | After electroacupuncture(Day 7)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
p300 cortical response wave latency | 7 days after electroacupuncture(Day 14)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.
p300 cortical response wave amplitude | 7 days after electroacupuncture(Day 14)
  An audiologist places small earphones in the ears and electrodes near the ears and on the forehead. Clicking sounds and tones go through the earphones, and electrodes measure how the hearing nerves and brain respond to the sounds.

CONTACTS AND LOCATIONS:
Overall Officials: China Medical University, Study Chair — China Medical University, China
Locations (1):
- China Medical University, Taichung, Taiwan